CLINICAL TRIAL: NCT02291887
Title: Genetic Analysis of Patients With Neovascular Age-Related Macular Degeneration Responsive to Ranibizumab But Resistant to Aflibercept
Brief Title: Genetic Analysis of Patients Responsive to Ranibizumab But Resistant to Aflibercept
Status: Completed | Type: Observational
Sponsor: Associated Retinal Consultants, Michigan (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ARCMichigan
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood from each patient will be drawn for genetic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neovascular ARMD Patients: Patients with Neovascular Age-Related Macular Degeneration Responsive to Ranibizumab but Resistant to Aflibercept Treatment
  Interventions: Drug: Ranibizumab; Drug: Aflibercept

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection of Ranibizumab
  Other Names: Lucentis
Drug: Aflibercept — Intravitreal injection of Aflibercept
  Other Names: Eylea

SUMMARY:
A cohort of patients responsive to treatment with ranibizumab but resistant to

aflibercept were identified in a previously conducted retrospective study. Identified

patients will have their blood drawn for genome wide sequencing. The sequencing

data will be compiled and analyzed in an attempt to identify a common genetic basis

for patients susceptible to ranibizumab but resistant to aflibercept.

DETAILED DESCRIPTION:
A cohort of patients responsive to treatment with ranibizumab but resistant to

aflibercept were identified in a previously conducted retrospective study. Identified

patients will have their blood drawn for genome wide sequencing. The sequencing

data will be compiled and analyzed in an attempt to identify a common genetic basis

for patients susceptible to ranibizumab but resistant to aflibercept.

Blood samples will be drawn for genetic analysis for all patients enrolled in the study.

The sample (1 tube- 6mL of blood) will be collected using - 8.5mL PAXgene Blood DNA

Tubes (http://www.qiagen.com/products/catalog/sample-technologies/dna-sample-

technologies/genomic-dna/paxgene-blood-dna-tubes).

Samples will be stored at -80 until time for analysis. Note that some blood draws will be performed at

satellite clinics and transported to main facility for storage in -80 freezer. It is the understanding of

ARC PI and staff that the PAXgene Blood DNA Tubes keep samples stable at room temp for 1-2

days.

However, staff will transport samples in timely fashion (room temp, on ice, dry ice,

etc), to -80 freezer for storage until all samples are collected. Once all samples are

collected, they will be shipped to Genentech for analysis. DNA extraction, the generation of genetic

data, and subsequent analysis will be performed at Genentech or via third party. DNA will be assayed

for polymorphisms through genome wide SNP chip or whole genome sequencing. The subject's

genotype or haplotype will be correlated with their visual response and OCT response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:

  * Demonstrate worsening of exudation when switched from ranibizumab to aflibercept
  * Ability to provide written informed consent and comply with study assessments for the full duration of the study

Exclusion Criteria:

* Any other condition that the investigator believes would pose a significant hazard to the subject

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 17 subjects from approximately 1 site in the United States will be enrolled. Eligible subjects will be administered and provided with a copy of informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Genetic characteristics of patients responsive to Ranibizumab but Resistant to Aflibercept | 1 day
  To determine a genetic basis for patients responsive to ranibizumab but resistant to aflibercept.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Wolfe, MD, MS, Principal Investigator — Associated Retinal Consultants
Locations (1):
- Associated Retinal Consultants, Royal Oak, Michigan, United States

REFERENCES:
- [Result] Eyetech Study Group. Anti-vascular endothelial growth factor therapy for subfoveal choroidal neovascularization secondary to age-related macular degeneration: phase II study results. Ophthalmology. 2003 May;110(5):979-86. doi: 10.1016/S0161-6420(03)00085-X. PMID 12750101
- [Result] Rosenfeld PJ, Rich RM, Lalwani GA. Ranibizumab: Phase III clinical trial results. Ophthalmol Clin North Am. 2006 Sep;19(3):361-72. doi: 10.1016/j.ohc.2006.05.009. PMID 16935211
- [Result] Michels S, Schmidt-Erfurth U, Rosenfeld PJ. Promising new treatments for neovascular age-related macular degeneration. Expert Opin Investig Drugs. 2006 Jul;15(7):779-93. doi: 10.1517/13543784.15.7.779. PMID 16787141
- [Result] Rosenfeld PJ, Heier JS, Hantsbarger G, Shams N. Tolerability and efficacy of multiple escalating doses of ranibizumab (Lucentis) for neovascular age-related macular degeneration. Ophthalmology. 2006 Apr;113(4):623.e1. doi: 10.1016/j.ophtha.2006.01.027. PMID 16581423
- [Result] Heier JS, Antoszyk AN, Pavan PR, Leff SR, Rosenfeld PJ, Ciulla TA, Dreyer RF, Gentile RC, Sy JP, Hantsbarger G, Shams N. Ranibizumab for treatment of neovascular age-related macular degeneration: a phase I/II multicenter, controlled, multidose study. Ophthalmology. 2006 Apr;113(4):633.e1-4. doi: 10.1016/j.ophtha.2005.10.052. Epub 2006 Feb 14. PMID 16483659
- [Result] Feigl B, Brown B, Lovie-Kitchin J, Lee L. Dynamics of retinal function after multiple photodynamic therapies in age-related macular degeneration: a report of cases. Doc Ophthalmol. 2005 Nov;111(3):135-48. doi: 10.1007/s10633-005-5319-7. Epub 2006 Mar 6. PMID 16523231
- [Result] D'Amico DJ. Diseases of the retina. N Engl J Med. 1994 Jul 14;331(2):95-106. doi: 10.1056/NEJM199407143310207. No abstract available. PMID 8208273